CLINICAL TRIAL: NCT05177575
Title: Incidence of Chronic Pain After Thoracotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2438
Record Dates: First submitted 2021-12-16; First posted 2022-01-04 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain; Postoperative Pain, Acute; Postoperative Pain, Chronic; Thoracotomy
Keywords: Postoperative Pain; Postoperative Pain, Acute; Postoperative Pain, Chronic; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thoracotomy application — The chronic pain findings of the patients who underwent thoracotomy will be questioned at the postoperative 3rd and 6th months.

SUMMARY:
Thoracotomy is frequently performed in thoracic surgery. It is widely accepted that thoracotomy causes severe acute pain. Many factors such as postoperative analgesia treatment plan, operation time, number of chest tubes, and duration of chest tube stay can affect acute pain. This acute pain prolongs the discharge time of the patients and increases the frequency of postoperative pulmonary complications and postoperative morbidity. Postoperative acute pain may cause chronic thoracotomy pain in the later period, and may adversely affect the quality of life of the patients.

This study aims to analyze the symptoms of chronic pain in the 3rd and 6th months postoperatively in patients who had undergone thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index (BMI) between 18-35 kg/m2
* Patients undergoing elective thoracotomy

Exclusion Criteria:

* Advanced cancer
* History of chronic analgesic therapy
* Patients with previous thoracic surgery
* Patients who were operated under emergency conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 years, in the ASA I-II-III risk group, with a BMI between 18-35 kg/m2 and undergoing thoracotomy will be included in the study.
  Patients under the age of 18 years and over the age of 65 years, with an ASA score of IV and above, with a BMI below 18 kg/m2 and above 35 kg/m2, who were operated under emergency conditions, and who received chronic pain treatment will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-03-16 (Estimated); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
Chronic pain symptoms at 3rd months. | Chronic pain symptoms at 3rd months.
  Chronic pain symptoms will be assessed using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Neuropathic pain symptoms (burning, stabbing, electric shock-like pain, tingling, numbness, pins, and needles feeling, hyperalgesia, allodynia, and hypoesthesia) will also be asked to the patients in the 3rd month after surgery.
Chronic pain symptoms at 6th months. | Chronic pain symptoms at 6th months.
  Chronic pain symptoms will be assessed using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Neuropathic pain symptoms (burning, stabbing, electric shock-like pain, tingling, numbness, pins, and needles feeling, hyperalgesia, allodynia, and hypoesthesia) will also be asked to the patients in the 6th month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No